CLINICAL TRIAL: NCT06422234
Title: Effect of Exergame-Based Exercise on Hamstring and Quadriceps Isokinetic Muscle Parameters, Balance and Explosive Power
Brief Title: Effect of Exergame-Based Exercise on Hamstring and Quadriceps Isokinetic Muscle Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACetinkaya001
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Exergaming; Sedentary Behavior; Muscle Strength
Keywords: Exergaming; Muscle Strength Dynamometer; Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exergame Group (Experimental): Participants will exercise 3 days a week for 6 weeks with the Ring Fit Adventure game on Nintendo Switch. The exergames to be played are selected by the physiotherapist and become more difficult as the weeks progress.
  Interventions: Other: Exergame
- Game-free Exercise Group (Active Comparator): The games selected for the exergame group will be held in a real environment, without games, 3 days a week for 6 weeks.
  Interventions: Other: Game-free Exercise
- Control Group (No Intervention): Participants in this group will continue their normal life routines and the evaluations will be repeated 6 weeks after the first evaluation.

INTERVENTIONS:
Other: Exergame — Video-based game exercises will be performed 3 days a week for 6 weeks. Participants will be taught how to play the games before starting the game called Ring Fit Adventure, one of the Nintendo Switch games. Among the games within Ring Fit, games that aim to increase lower extremity muscle strength, core stabilization and balance have been selected, and game types and number of repetitions are changed every week.
  Arms: Exergame Group
Other: Game-free Exercise — All activities in the exergame group were done without games and screens. The progression of the exercises proceeds in the same way as the other group.
  Arms: Game-free Exercise Group

SUMMARY:
The aim of this study is to investigate the effects of two different exercise methods (video-based game exercise group and real (non-game) exercise group) to increase knee strength in healthy individuals on muscle strength, balance and lower extremity functional parameters. In our study, it will be revealed which technique will have what effect in the strengthening, which will be done by taking certain criteria into consideration. Participants will be randomized into three different groups. Two groups, except the control group, will exercise three times a week for 6 weeks. All participants will be assessment twice in total, at the beginning of the study and 6 weeks later. It is thought that the results obtained here will contribute to the literature.

DETAILED DESCRIPTION:
The study was planned to include individuals studying at Halic University, who met the inclusion criteria and volunteered to participate in the study. Evaluated participants will be randomly assigned to three different groups (control group, video-based game exercise group, real game-free exercise group). The sealed envelope method will be used in randomization. All evaluations by the same physiotherapist will be performed twice, before exercise and after 6 weeks of exercise. Both exercise groups will practice under the supervision of a physiotherapist. The control group will not exercise and will only be evaluated twice. At the end of the study, those in the control group will be able to participate in any exercise group they want for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 18-25
* Being a 1st or 2nd year physiotherapy and rehabilitation student or a student in any department other than sports sciences
* Being sedentary or underweight according to fit score
* Being at normal values according to body mass index
* Full knee flexion-extension joint range of motion
* Volunteering to participate in the study

Exclusion Criteria:

* Knee pain, history of injury in the last 6 months,
* Doing regular physical activity in the last 6 months,
* Neurological, cardiorespiratory, musculoskeletal, endocrine, renal, metabolic and other related disease(s) that will prevent the performance of exercises
* History of lower extremity orthopedic surgery
* Chronic use of medications or anti-inflammatory drugs

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Isokinetic Evaluation-Peak Torque | at baseline and at week 6
  Biodex System 4 device will be used to evaluate quadriceps and hamstring isokinetic muscle strength. All tests were planned to be performed on the dominant and non-dominant sides of the participants. Isokinetic muscle strength test will be performed in concentric/concentric mode at speeds of 60°/sec, 90°/sec, 240°/sec in concentric strength test. Isokinetic test will be performed at 0° extension and 90° flexion joint range of motion. Before the isokinetic test, the participant will have 2 repetitions at 60°/sec for adaptation, and then 5 repetitions for the test. After the participant rests for 120 seconds, the participant will first have 4 repetitions for adaptation and then 15 repetitions for the test at 240°/sec. During the tests, the participant will be verbally motivated by the same person. .As a result of the tests, quadriceps and hamstring peak torque (PT) values will be recorded.
Isokinetic Evaluation-Peak Torque / Body Weight | at baseline and at week 6
  Biodex System 4 device will be used to evaluate quadriceps and hamstring isokinetic muscle strength. All tests were planned to be performed on the dominant and non-dominant sides of the participants. Isokinetic muscle strength test will be performed in concentric/concentric mode at speeds of 60°/sec, 90°/sec, 240°/sec in concentric strength test. Isokinetic test will be performed at 0° extension and 90° flexion joint range of motion. Before the isokinetic test, the participant will have 2 repetitions at 60°/sec for adaptation, and then 5 repetitions for the test. After the participant rests for 120 seconds, the participant will first have 4 repetitions for adaptation and then 15 repetitions for the test at 240°/sec. During the tests, the participant will be verbally motivated by the same person. As a result of the tests, peak torque/body weight (PT/VA) values will be recorded.
Isokinetic Evaluation-Peak Torque / Hamstring/Quadriceps (H/Q) | at baseline and at week 6
  Biodex System 4 device will be used to evaluate quadriceps and hamstring isokinetic muscle strength. All tests were planned to be performed on the dominant and non-dominant sides of the participants. Isokinetic muscle strength test will be performed in concentric/concentric mode at speeds of 60°/sec, 90°/sec, 240°/sec in concentric strength test. Isokinetic test will be performed at 0° extension and 90° flexion joint range of motion. Before the isokinetic test, the participant will have 2 repetitions at 60°/sec for adaptation, and then 5 repetitions for the test. After the participant rests for 120 seconds, the participant will first have 4 repetitions for adaptation and then 15 repetitions for the test at 240°/sec. During the tests, the participant will be verbally motivated by the same person. As a result of the tests, Hamstring/Quadriceps (H/Q) values will be recorded.
Isokinetic Evaluation-Peak Torque / Total Work | at baseline and at week 6
  Biodex System 4 device will be used to evaluate quadriceps and hamstring isokinetic muscle strength. All tests were planned to be performed on the dominant and non-dominant sides of the participants. Isokinetic muscle strength test will be performed in concentric/concentric mode at speeds of 60°/sec, 90°/sec, 240°/sec in concentric strength test. Isokinetic test will be performed at 0° extension and 90° flexion joint range of motion. Before the isokinetic test, the participant will have 2 repetitions at 60°/sec for adaptation, and then 5 repetitions for the test. After the participant rests for 120 seconds, the participant will first have 4 repetitions for adaptation and then 15 repetitions for the test at 240°/sec. During the tests, the participant will be verbally motivated by the same person. As a result of the tests, total work values will be recorded.

SECONDARY OUTCOMES:
Proprioception Assessment | at baseline and at week 6
  Individuals' joint position sense of the knee joint will be evaluated at 30°, 45° and 75° knee flexion angles using the Biodex System 4 device. While the individual's eyes are closed, the knee joint will be brought to the targeted angle by the researcher, and the subject will be asked to stay in this position for 5 seconds and perceive this angular position. Afterwards, the individuals' knee angle will be flexed to 90° and they will be asked to bring the knee joint to the targeted angle. The test will be repeated three times and the average of the deviation degrees from the targeted angle in the three tests will be recorded regardless of the direction of movement. The less deviation from the target angle, the better the sense of proprioception.
Vertical Jump Test | at baseline and at week 6
  It is asked to jump to maximum height from the double-leg squat position. Between jumps, 15 to 30 seconds of listening time is given for recovery. Athletes are asked to perform 3 repetitions and the average of the values is recorded. The jump height is recorded in centimeters. The EZEJUMP (vertical jump testing system) System will be used for this test.The higher the jump height, the better the performance.
Standing long jump | at baseline and at week 6
  It is asked to open his legs shoulder-width apart, and without taking a step, he jumps forward, gaining momentum with his arms. The distance between the starting line and the heel closest to this line is recorded as the score. The jump distance is recorded in centimeters Three attempts are made and the best score is noted. The higher the jump distance, the better the performance.
Flamingo Balance Test | at baseline and at week 6
  While the individual tries to balance on a 15 cm long, 4 cm wide wooden plate prepared in the dimensions specified in the literature, the number of times he falls in 1 minute will be recorded. He stands on the bench with his dominant foot lengthwise, bends his free foot backwards and holds it with his hand on the same side. The other arm is released to maintain balance. During this period, the stopwatch will be stopped during each fall and the individual will be waited to get into position again. As the number of falls decreases during one minute, static balance performance increases.
Modified Star Balance Test | at baseline and at week 6
  The maximum distance that a person can travel while balancing on one leg in three directions is recorded in centimeters. At the furthest point they lie down, the person is asked to lightly touch the ground and balance standing again. The test is completed by moving clockwise or counterclockwise. While stretching, your hands are asked to be on the iliac crests. A trial tour is conducted before the test. The average of the subject's three attempts in each direction is taken, the result is divided by the leg length and multiplied by 100. Increasing the distance a person can reach with the other leg while remaining in balance indicates that dynamic balance performance increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Çetinkaya, MSc, Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Eyüpsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No